CLINICAL TRIAL: NCT02464722
Title: Comparision Between Hemodynamic Response of Dexmedetomidine and Remifentanil for Epinephrine Local Injection in Patient With Endoscopic Sinus Surgery Under General Anesthesia
Brief Title: Comparision Between Hemodynamic Response of Dexmedetomidine and Remifentanil on Anesthesia in Endoscopic Sinus Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Joonchul Jang, Resident, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ED15010
Record Dates: First submitted 2015-05-27; First posted 2015-06-08 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Hemodynamic Instability
Keywords: Remifentanil; Dexmedetomidine; Endoscopic sinus surgery
MeSH Terms: interventions — Dexmedetomidine; Remifentanil; Epinephrine; Propofol; Rocuronium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine (Experimental): 1. Before induction of Anesthesia, 1 mcg/kg iv loading dose of dexmedetomidine over 10 minutes.
  2. Anesthesia was induced with propofol 2 mg kg-1 , rocuronium 0.6 mg kg-1
  3. After Mask ventilation with 6 vol% desflurane in 100% oxygen for 3 minutes, tracheal intubation was done
  4. Later, an infusion was started at the rate of 0.4-0.8mcg/kg/min. The infusion rate was adjusted according to the patient's response, to achieve a mean arterial pressure between 60 and 80 mmHg.
  5. Before the start of surgery, 1/100000 epinephrine infiltration was administered to the nasal passages by the surgeon.
  6. At the end of surgery, discontinuation of desflurane and dexmedetomidine, sending recovery room.
  Interventions: Drug: Dexmedetomidine; Drug: Epinephrine; Drug: Propofol; Drug: Rocuronium
- Remifentanil (Active Comparator): 1. Anesthesia was induced with propofol 2 mg kg-1 , rocuronium 0.6 mg kg-1
  2. Mask ventilation with 6 vol% desflurane in 100% oxygen for 2 minutes.
  3. After 1 mcg/kg iv loading dose of remifentanil over a period of 1 minutes. tracheal intubation was done.
  4. Later, an infusion was started at the rate of 0.2-0.4mcg/kg/min. The infusion rate was adjusted according to the patient's response, to achieve a mean arterial pressure between 60 and 80 mmHg.
  5. Before the start of surgery, 1/100000 epinephrine infiltration was administered to the nasal passages by the surgeon.
  6. At the end of surgery, discontinuation of desflurane and remifentanil, sending recovery room.
  Interventions: Drug: Remifentanil; Drug: Epinephrine; Drug: Propofol; Drug: Rocuronium

INTERVENTIONS:
Drug: Dexmedetomidine — 1 mcg/kg iv loading dose of remifentanil over a period of 60 seconds. Later, an infusion was started at the rate of 0.2-0.4mcg/kg/min.
  Other Names: dexmedetomidine hydrochloride
  Arms: Dexmedetomidine
Drug: Remifentanil — 1 mcg/kg iv loading dose of remifentanil over a period of 10 minutes. Later, an infusion was started at the rate of 0.4-0.8mcg/kg/min.
  Other Names: remifentanil hydrochloride
  Arms: Remifentanil
Drug: Epinephrine — Before the start of surgery, 1/100000 epinephrine infiltration was administered to the nasal passages by the surgeon.
Drug: Propofol — Anesthesia was induced with propofol 2 mg kg-1
Drug: Rocuronium — Anesthesia was induced with rocuronium 0.6 mg kg-1

SUMMARY:
During endoscopic sinus surgery (ESS), epinephrine local injection and controlled hypotension is essential in order to increase the visibility in the operative field and reduce the risk. This study is comparing of dexmedetomidine and remifentanil before epinephrine local injection for controlled hypotension during ESS.

DETAILED DESCRIPTION:
During endoscopic sinus surgery (ESS), epinephrine local injection and controlled hypotension is essential in order to increase the visibility in the operative field and reduce the risk.

Epinephrine local injection and controlled hypotensive anesthesia is commonly used in several surgical interventions using different techniques. However, choosing the ideal agent is still a controversial topic.

In the current study, the effects and safety of remifentanil, which is an μ opioid receptor agonist and dexmedetomidine, an α-2 agonist; when used before epinephrine local injection for controlled hypotension in ESS, are compared.

After obtaining Institutional Review Board approval and written informed consent, 40 patients is enrolling in this study.

Participants is divided by two groups randomly as the Dexmedetomidine group and the Remifentanil group.

A correctly sized facemask and 100 % oxygen was used for pre-oxygenation. General anesthesia was induced with iv Propofol 1.5-2 mg kg-1. Endotracheal intubation was performed with the aid of iv Rocuronium 0.6 kg-1. Ventilation was controlled with 50% air in oxygen to maintain end-tidal carbon dioxide pressure at 30-36 mmHg. Desflurane was used for maintenance.

Before epinephrine injection, In group Remifentanil, Participants received 1 mcg kg-1 iv loading dose of remifentanil over a period of 60 seconds. Later, an infusion was started at the rate of 0.2-0.4 mcg kg-1 h-1. The infusion rate was adjusted according to the Participants response, to achieve a mean arterial pressure between 60 and 75 mmHg. In group Dexmedetomidine, patients received a 1 mcg kg-1 loading dosage of dexmedetomidine within 10 min and later, infusion was started at the rate of 0.4-0.8 mcg kg-1min-1. The infusions began before tracheal intubation in both groups. Standard dose epinephrine local infiltration was administered to the nasal passages by the surgeon.

Systolic Arterial Pressure,Diastolic Arterial Pressure,Mean arterial blood pressure, Heart Rate were recorded every 5min, from the beginning of anesthesia and every 1min, from the epinephrine local injection. Perioperative hypotension and bradycardia were defined as mean arterial blood pressure < 50 mmHg or 50 beat/min respectively. Ephedine was administered intravenously for the treatment of hypotension. Atropine 0.5 mg was administered intravenously for the treatment of bradycardia.

All infusions were stopped 5 min before the end of surgery. After surgery, the surgeon evaluated the dryness of the surgical area. Recovery time was recorded in the postoperative period. An investigators employing the Modified Observer's Assessment of Alertness/Sedation Scale assessed recovery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist[ASA] class 1-2
* scheduled Endoscopic sinus surgery
* written informed consent

Exclusion Criteria:

* allergy of opioids, neuromuscular blocking drugs or other medications used during general anesthesia
* known or suspected upper respiratory infection
* suspected difficult tracheal intubation
* Uncontrolled Hypertension
* known or suspected psychologic disorder
* known or suspected significant renal dysfunction
* known or suspected severe hepatic dysfunction
* known or suspected significant cardiovascular dysfunction

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-08; Primary Completion 2015-11 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Change in blood pressure | At the time from epinephrine local injection (1,2,3,4,5,6,7,8,9,10,11,12,13,14,15 minutes)

SECONDARY OUTCOMES:
Conditions during Surgery | At the time during Surgery
  We assessed conditions during ESS(Surgeon evaluated the dryness of the surgical area using six point quality scale.)

OTHER OUTCOMES:
Change in heart rate | At the time from epinephrine local injection (1,2,3,4,5,6,7,8,9,10,11,12,13,14,15 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Jangeun Cho, M.D, Ph.D, Principal Investigator — Anesthesia and Pain medicine department, Korea University Anam Hospital

REFERENCES:
- [Result] Lee J, Kim Y, Park C, Jeon Y, Kim D, Joo J, Kang H. Comparison between dexmedetomidine and remifentanil for controlled hypotension and recovery in endoscopic sinus surgery. Ann Otol Rhinol Laryngol. 2013 Jul;122(7):421-6. doi: 10.1177/000348941312200702. PMID 23951692